CLINICAL TRIAL: NCT03543657
Title: A Randomized, Active-controlled, Double-blinded, Double-dummy, Parallel-group, Multicenter Study to Investigate the Efficacy and Safety of Oral Molidustat in Comparison to Darbepoetin Alfa in Dialysis Subjects Treated With Erythropoiesis-Stimulating Agents (ESAs)
Brief Title: Maintenance Treatment of Renal Anemia in Dialysis Subjects
Acronym: MIYABI HD-M
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19352
Record Dates: First submitted 2018-05-22; First posted 2018-06-01 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Anemia; Renal Insufficiency, Chronic
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — molidustat; Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Molidustat group (Experimental): Subjects in the molidustat group will receive molidustat and darbepoetin alfa placebo.
  Interventions: Drug: Molidustat (BAY85-3934); Drug: Placebo of Darbepoetin alfa
- Darbepoetin alfa group (Active Comparator): Subjects in the darbepoetin alfa group will receive molidustat placebo and darbepoetin alfa.
  Interventions: Drug: Darbepoetin alfa; Drug: Placebo of Molidustat (BAY85-3934)

INTERVENTIONS:
Drug: Molidustat (BAY85-3934) — Starting dose of molidustat will be titrated based on the subject's Hb (Hemoglobin) response. Administrated orally once daily (OD).
  Arms: Molidustat group
Drug: Darbepoetin alfa — Starting dose of darbepoetin alfa will be titrated based on the subject's Hb (Hemoglobin) response. Administrated weekly or once every two weeks by intravenous injection.
  Arms: Darbepoetin alfa group
Drug: Placebo of Molidustat (BAY85-3934) — Matching placebo of Molidustat.
  Arms: Darbepoetin alfa group
Drug: Placebo of Darbepoetin alfa — Matching placebo of Darbepoetin alfa.
  Arms: Molidustat group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of molidustat in comparison to darbepoetin alfa in dialysis subjects with renal anemia who are treated with Erythropoiesis-Stimulating Agents (ESAs).

ELIGIBILITY:
Inclusion Criteria:

* Subject with ESKD (end-stage kidney disease) on regular dialysis (including, hemodiafiltration, hemofiltration, hemodialysis, and other modalities except for peritoneal dialysis) weekly or more than weekly for at least 12 weeks prior to randomization
* Body weight (after dialysis) > 40 and ≤ 160 kg at screening
* Male or female subject ≥ 20 years of age at screening
* At least one kidney
* Treated with weekly or bi-weekly dose of darbepoetin alfa, monthly or bi-weekly dose of epoetin beta pegol, OR weekly, biweekly, twice or three times per week dose of epoetin alfa/beta, and having had no more than one dose change within 8 weeks prior to randomization
* Mean screening Hb level ≥ 9.5 and < 12.0 g/dL (mean of all central laboratory Hb levels before dialysis [at least 2 measurements must be taken ≥ 2 days apart] during the screening period, AND all Hb level must be measured by the central laboratory, AND the difference between the lowest level and highest level is < 1.2 g/dL), with the last screening Hb level measurement within 14 days prior to randomization
* Ferritin ≥ 100 ng/mL or transferrin saturation ≥ 20% at screening
* Serum folate level and serum vitamin B12 level above lower limit of normal (LLN) at screening

Exclusion Criteria:

* New York Heart Association (NYHA) Class III or IV congestive heart failure
* History of cardio- (cerebro-) vascular events (e.g., unstable angina, myocardial infarction, stroke, pulmonary thromboembolism, and acute limb ischemia) within 6 months prior to randomization
* Sustained, poorly controlled arterial hypertension (defined as systolic BP (blood pressure) ≥ 180mmHg or diastolic BP ≥ 110mmHg) or hypotension (defined as systolic BP < 90mmHg) at randomization
* Proliferative choroidal or retinal disease, such as neovascular agerelated macular degeneration or proliferative diabetic retinopathy requiring invasive treatment (e.g., intraocular injections or laser photocoagulation) at screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2018-06-23 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
The mean Hb level during the evaluation period | From week 33 to 36
The change in mean Hb level during the evaluation period from baseline | Baseline and week 33 to 36

SECONDARY OUTCOMES:
Responder rate: proportion of responders among the subjects | From week 33 to 36
  Responder is defined as meeting all of the following criteria:
  (i) Mean of the Hb levels in the target range (ii) ≥ 50% of the Hb levels in the target range (iii) No rescue treatment
Proportion of subjects who meet each component of the response | From week 33 to 36
  Response:
  (i) Mean of the Hb levels in the target range (ii) ≥ 50% of the Hb levels in the target range (iii) No rescue treatment
Hb level | Up to 52 weeks
Change in Hb level | Baseline and up to 52 weeks
Proportion of subjects whose mean hemoglobin level is in the target range | From week 33 to 36
Proportion of subjects whose mean hemoglobin level is above the target range | From week 33 to 36
Proportion of subjects whose mean hemoglobin level is below the target range | From week 33 to 36
Proportion of subjects with hemoglobin levels in the target range | Up to 52 weeks
Proportion of subjects with hemoglobin levels above the target range | Up to 52 weeks
Proportion of subjects with hemoglobin levels below the target range | Up to 52 weeks
Proportion of subjects whose maximum rise in Hb between each consecutive visits is above 0.5 g/dL/week | Up to 52 weeks
  Defined as change in Hb level / duration between two visits (weeks)
Number of participants with serious adverse events | Up to 52 weeks
Maximum concentration (Cmax) | At baseline, week 8, week 24 and week 52
Area under the concentration-time curve (AUC) | At baseline, week 8, week 24 and week 52
EPO (Erythropoietin) serum concentration | At baseline, week 8, week 24 and week 52

CONTACTS AND LOCATIONS:
Locations (53):
- Japan (53):
  - Hakuyoukai Medical corporation Hakuyoukai Hospital, Nagoya, Aichi-ken
  - Shinkashiwa Clinic, Kashiwa, Chiba
  - Kisarazu Clinic, Kisarazu, Chiba
  - Kuwajima Clinic, Niihama, Ehime
  - Sabae kidney Clinic, Sabae, Fukui
  - Houshikai Kano hospital, Kasuya-gun, Fukuoka
  - Saiseikai Yahata General Hospital, Kitakyushu, Fukuoka
  - Sanshikai Toho Hospital, Midori, Gunma
  - Asahikawa-Kosei General Hospital, Asahikawa, Hokkaido
  - Koizumi Cardiology Medical Clinic, Chitose, Hokkaido
  - Ishikari Hospital, Ishikari, Hokkaido
  - Itami Kidney Clinic, Noboribetsu, Hokkaido
  - Souen Central Hospital, Sapporo, Hokkaido
  - Ibaraki Prefectural Central Hospital, Kasama, Ibaraki
  - Japanese Red Cross Koga Hospital, Koga, Ibaraki
  - Mito Kyodo General Hospital, Mito, Ibaraki
  - Tokiwa Clinic, Totte, Ibaraki
  - Tsuchiura Beryl Clinic, Tsuchiura, Ibaraki
  - Kikuchi Medical Clinic, Tsukuba, Ibaraki
  - Public Central Hospital of Matto Ishikawa, Hakusan, Ishikawa-ken
  - Kaisei Hospital, Sakaidechō, Kagawa-ken
  - Honatsugi Medical Clinic, Atsugi, Kanagawa
  - Chigasaki Central Clinic, Chigasaki, Kanagawa
  - Toshiba Rinkan Hospital, Sagamihara, Kanagawa
  - Yokohama Jin Clinic, Yokohama, Kanagawa
  - Eda Clinic, Yokohama, Kanagawa
  - Kaminagaya Saitou Clinic, Yokohama, Kanagawa
  - Seisuikai Yoshioka Mahoroba Clinic, Kurokawa-gun, Miyagi
  - Eijinkai Hospital, Ōsaki, Miyagi
  - Iida Hospital, Iida, Nagano
  - Kanno Dialysis & Vascular Access Clinic, Matsumoto, Nagano
  - Matsumoto City Hospital, Matsumoto, Nagano
  - Maruko Central Hospital, Ueda, Nagano
  - Arisawa General Hospital, Hirakata, Osaka
  - Toyonaka Keijinkai Clinic, Toyonaka, Osaka
  - Hanyu General Hospital, Hanyū, Saitama
  - Higashimatsuyamakohjin Clinic, Higashi-Matsuyama, Saitama
  - Saiyu Clinic, Koshigaya, Saitama
  - Todachuo General Hospital, Toda, Saitama
  - Hachioji Azumacho Clinic, Hachiōji, Tokyo
  - Kodaira Kitaguchi Clinic, Kodaira, Tokyo
  - Saint Hill Hospital, Ube, Yamaguchi
  - Medical corporation association Shunshin-kai Inage hospital, Chiba
  - Ikeda Vascular Access Nephrology Dialysis, Fukuoka
  - Oohashi internal medicine circulatory Clinic, Fukuoka
  - Ueki Imafuji Clinic, Kumamoto
  - Medical Corporation Suzukihinyoukika, Nagano
  - Nagasaki Kidney Hospital, Nagasaki
  - Akagaki Clinic, Osaka
  - Nishi Shinryosho, Osaka
  - Chibune Clinic, Osaka
  - Iwatsuki-minami Hospital, Saitama
  - Yamagata Tokushukai Hospital, Yamagata

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Akizawa T, Taguchi M, Matsuda Y, Iekushi K, Yamada T, Yamamoto H. Molidustat for the treatment of renal anaemia in patients with dialysis-dependent chronic kidney disease: design and rationale of three phase III studies. BMJ Open. 2019 Jun 14;9(6):e026602. doi: 10.1136/bmjopen-2018-026602. PMID 31203241
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/